CLINICAL TRIAL: NCT05725538
Title: Efficacy of Exercise-based mHealth Intervention for Patients With Post-acute COVID-19 Syndrome Based on Fatigue, Fitness, Post-exertional Dyspnea, Pain, Anxiety, Depression, Cognitive Function, and Quality of Life: a Randomized Clinical Trial.
Brief Title: Exercise Intervention Using mHealth in Patients With Post-Acute COVID-19 Syndrome: a Randomized Clinical Trial
Acronym: COVIDReApp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Jose A. Moral-Munoz, Assistant Professor, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVIDReApp
Record Dates: First submitted 2023-02-07; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Post-Acute COVID19 Syndrome; Long COVID; Post COVID-19 Condition
Keywords: smartphone; mHealth; mobile health; telerehabilitation; exercise; Post-Acute COVID-19 Syndrome; Long COVID; Post-COVID Condition; COVIDReApp
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A single-blind method will be carried out on the persons collecting and analysing the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVIDReApp Group (Experimental): The intervention group will complete a program of exercise guided by a m-health system (COVIDReApp) for 24 weeks.
  Interventions: Device: COVIDReApp Group
- Control Group (Active Comparator): The comparator group will complete a program of exercise in a traditional way (exercises will be provided in paper format) for 24 weeks.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: COVIDReApp Group — The COVIDReApp group will be required to complete an exercise program guided by an m-health system for three times per week during 24 weeks. A 60-minute program, following the recommendations of the American College of Sports Medicine. The daily session will be divided into:
  * Warm-up: 5 min. walking so that the patient can hold a conversation , monopodial balance exercise, core exercise and other respiratory and joint mobility exercises.
  * Aerobic training: Walking for 10 to 20 min. so that the patient can maintain a conversation, but having to stop to breathe from time to time.
  * Strengthening: It will focus on 7 exercises. a) squats, b) dead weight with stiff legs, c) lateral pull-ups, d) inverted flies, e) flies, f) unilateral rowing and g) lateral raises.
  * Cool down: It will consist of stretching exercises. a) shoulders, b) triceps, c) chest, d) quadriceps, e) hamstrings, and f) back.
  Arms: COVIDReApp Group
Other: Control Group — Participants will receive the same intervention in the traditional way, they will receive the exercise program in paper format. They will receive a document with photos and descriptions of the exercises to be performed. Their doctors will determine if the patients will be able to exercise regularly and they will perform them for 24 weeks.
  Arms: Control Group

SUMMARY:
Post-Acute Syndrome COVID-19 is a disease resulting from infection by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). It is estimated that between 10 and 35% of infected persons suffer symptoms afterwards, and in hospitalized patients it can reach 85%. These sequelae have individual, social and economic repercussions, so effective rehabilitation alternatives are necessary. Physical exercise is recommended as rehabilitation for these patients. Moreover, the implementation of m-Health supported interventions is a proven alternative in patients with Post-Acute COVID-19 Syndrome or other conditions, which improves therapeutic adherence and patient autonomy. Therefore, the development and evaluation of the effectiveness of an exercise-based m-Health system for application in patients with Post-Acute COVID-19 Syndrome responds to a need.

Our hypothesis is that a mobile health technology based on physical exercise recommendations for patients with Post-Acute COVID-19 Syndrome will improve fatigue, physical fitness, post-exertional dyspnea, pain intensity, anxiety, depression, cognitive function, and quality of life. Therefore, this project aims to evaluate the efficacy of the mobile health technology system (COVIDReApp) based on physical exercise recommendations for patients with COVID-19 Post-Acute Syndrome based on its results on fatigue, physical condition, post-exertional dyspnea, pain intensity, anxiety and depression, cognitive function and quality of life.

The achievement of the present project will serve to analyze the benefits of a physical exercise program in patients with COVID-19 Post-Acute Syndrome and identify those patients in whom the benefits will be greatest and whose implementation will have the highest priority.

ELIGIBILITY:
Eligible participants will be patients who have had COVID-19 at any time since the onset of the pandemic and even have Acute Post-CoVID-19 Syndrome, identified by their physicians and recruited from routine outpatient appointments at the Post-CoVID-19 Service of the Hospital Universitario Puerta del Mar, Cadiz, Spain.

Their physicians will give them an appointment for a future session in which potential participants will be provided with patient information and the consent form, and will be contacted approximately 48 hours later to discuss their willingness to participate.

Inclusion Criteria:

* Male and female patients.
* Over 18 years of age.
* Absence of cognitive and physical deficits that would preclude physical exercise.
* Owner of a smartphone with Internet access.
* Ability to understand and write in Spanish.

Exclusion criteria:

* Concomitant diseases that prevent physical exercise.
* Contraindications to physical exercise detected by physicians.
* Participation in moderate-intensity activities (more than 30 minutes and 3 times per week) at the time of study initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Longitudinal Change from Baseline up to 24 Weeks Follow-up in Fatigue (Fatigue Severity Scale (FSS)) | Baseline, 4 weeks post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.
  The FSS consists of 9 items related to the interference of fatigue with specific activities and rates the perceived severity of fatigue on a 7-point scale (1 = "strongly disagree"; 7 = "strongly agree").
Longitudinal Change from Baseline up to 24 Weeks Follow-up in Post-exertional dyspnoea (Dyspnoea-12) | Baseline, 4 weeks post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.
  Post-exertional dyspnea is assessed using the Dyspnea-12, a short questionnaire that takes into account both sensory and affective factors that may play a role in dyspnea. Each item in the questionnaire is scored from 0, if the symptom is mild, to 3, if it is severe, and the total score is the sum of the scores for all items. Six of the questions relate to sensory aspects and 6 to affective aspects of dyspnea. The total score ranges from 0 to 36, with 36 being the highest possible severity and 0 being the lowest.
Longitudinal Change from Baseline up to 24 Weeks Follow-up in Quality of life (SF-12v2) | Baseline, 4 weeks post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.
  The Short Form-12 (SF-12v2) will be administered to assess quality of life. This instrument contains 12 items that allow us to calculate the profile of 8 dimensions: (physical functioning, role-physical, bodily pain, general health perception, vitality, social functioning, role-emotional, and mental health) and two global scores: the physical health (PCS-12) and the mental health (MCS-12) component summary. Each global score ranges from 0 to 100, with higher scores indicating better health.

SECONDARY OUTCOMES:
Longitudinal Change from Baseline up to 24 Weeks Follow-up in Pain intensity (Visual Analog Scale (VAS)) | Baseline, 4 weeks post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.
  VAS is a scale used to rate the patient's pain intensity. The patient chooses a number from 0 to 10 (11-point numeric scale) that represents the best level of pain that the patient can imagine. A score of 0 represents no pain and 10 represents the worst pain imaginable.
Longitudinal Change from Baseline up to 24 Weeks Follow-up in Upper limb strength (Arm curl test) | Baseline, 4 weeks post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.
  The Arm Curl Test assesses upper body strength by determining the number of times a hand weight (2.3 kg) can be curled through a full range of motion in 30 seconds.
Longitudinal Change from Baseline up to 24 Weeks Follow-up in Lower limb strength (Chair stand test) | Baseline, 4 weeks post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.
  The chair stand test evaluates lower body muscular strength by counting the number of times a person can go from a sitting position to a standing position in 30 seconds.
Longitudinal Change from Baseline up to 24 Weeks Follow-up in Functional capacity and endurance (Two-minute walk test (2MWT)) | Baseline, 4 weeks post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.
  The two-minute walk test (2MWT) assesses walking ability, functional endurance and functional capacity. It consists of measuring the distance the patient can walk for 2 minutes as fast as he or she can safely without assistance.
Longitudinal Change from Baseline up to 24 Weeks Follow-up in Depression and/or anxiety (Hospital Anxiety and Depression Scale (HADs) | Baseline, 4 weeks post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.
  Depression and anxiety are assessed using the Hospital Anxiety and Depression Scale (HADS), which consists of 14 items divided into two subscales: anxiety (HADS-A) and depression (HADS-D).
Longitudinal Change from Baseline up to 24 Weeks Follow-up in Cognitive function (Test Your Memory (TYM)) | Baseline, 4 weeks post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.
  The Test Your Memory (TYM) screening test is used to assess cognitive function. This tool consists of 10 items with a total score ranging from 0 to 50, calculated on 10 cognitive dimensions: executive function, anterograde memory, visuospatial ability, naming, similarities, verbal fluency, calculation, retrograde memory, copying, orientation. The cut-off point is 42/50 (≤41 points indicates cognitive dysfunction) and a higher score indicates better cognitive performance.
Longitudinal Change from Baseline up to 24 Weeks Follow-up in Height, weight, and body mass index | Baseline, 4 weeks post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.
  Body measurements: height (standard height meter), weight, and body mass index (Tanita Model TBF-310 GS Weight Scale, Tanita Corporation of America, Inc., Arlington Heights, IL).
Baseline of sociodemographic variables | Baseline.
  A structured questionnaire will be used to collect sociodemographic data, including the following variables: gender, age, socioeconomic status, marital status, education level, employment status, clinical data, and use of alternative therapies.
Daily registry of the exercise difficulty (Borg Rating of Perceived Exertion Scale (RPE)) | Only CovidReApp group: Daily.
  CovidReApp system will register the daily exercise, which allows us to know the exercise difficulty of each exercise.
Daily registry of the adherence (CovidReApp log registration and self-reported) | Daily.
  The information is collected by the system only in the COVIDReApp group.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Puerta del Mar, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared with third parties.

REFERENCES:
- [Background] Soriano JB, Murthy S, Marshall JC, Relan P, Diaz JV; WHO Clinical Case Definition Working Group on Post-COVID-19 Condition. A clinical case definition of post-COVID-19 condition by a Delphi consensus. Lancet Infect Dis. 2022 Apr;22(4):e102-e107. doi: 10.1016/S1473-3099(21)00703-9. Epub 2021 Dec 21. PMID 34951953
- [Background] Lopez-Leon S, Wegman-Ostrosky T, Perelman C, Sepulveda R, Rebolledo PA, Cuapio A, Villapol S. More than 50 long-term effects of COVID-19: a systematic review and meta-analysis. Sci Rep. 2021 Aug 9;11(1):16144. doi: 10.1038/s41598-021-95565-8. PMID 34373540
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Raman B, Cassar MP, Tunnicliffe EM, Filippini N, Griffanti L, Alfaro-Almagro F, Okell T, Sheerin F, Xie C, Mahmod M, Mozes FE, Lewandowski AJ, Ohuma EO, Holdsworth D, Lamlum H, Woodman MJ, Krasopoulos C, Mills R, McConnell FAK, Wang C, Arthofer C, Lange FJ, Andersson J, Jenkinson M, Antoniades C, Channon KM, Shanmuganathan M, Ferreira VM, Piechnik SK, Klenerman P, Brightling C, Talbot NP, Petousi N, Rahman NM, Ho LP, Saunders K, Geddes JR, Harrison PJ, Pattinson K, Rowland MJ, Angus BJ, Gleeson F, Pavlides M, Koychev I, Miller KL, Mackay C, Jezzard P, Smith SM, Neubauer S. Medium-term effects of SARS-CoV-2 infection on multiple vital organs, exercise capacity, cognition, quality of life and mental health, post-hospital discharge. EClinicalMedicine. 2021 Jan 7;31:100683. doi: 10.1016/j.eclinm.2020.100683. eCollection 2021 Jan. PMID 33490928
- [Background] Leite VF, Rampim DB, Jorge VC, de Lima MDCC, Cezarino LG, da Rocha CN, Esper RB; Prevent Senior COVID-19 Rehabilitation Study. Persistent Symptoms and Disability After COVID-19 Hospitalization: Data From a Comprehensive Telerehabilitation Program. Arch Phys Med Rehabil. 2021 Jul;102(7):1308-1316. doi: 10.1016/j.apmr.2021.03.001. Epub 2021 Mar 10. PMID 33711279
- [Background] Ausin-Garcia C, Cervilla-Munoz E, Millan-Nunez-Cortes J. Long-term consequences of SARS-COV2 infection: Long-Covid patterns and possible public health implications. Med Clin (Barc). 2021 Oct 8;157(7):e293-e294. doi: 10.1016/j.medcli.2021.02.022. Epub 2021 May 6. No abstract available. PMID 34030861
- [Background] Curci C, Pisano F, Bonacci E, Camozzi DM, Ceravolo C, Bergonzi R, De Franceschi S, Moro P, Guarnieri R, Ferrillo M, Negrini F, de Sire A. Early rehabilitation in post-acute COVID-19 patients: data from an Italian COVID-19 Rehabilitation Unit and proposal of a treatment protocol. Eur J Phys Rehabil Med. 2020 Oct;56(5):633-641. doi: 10.23736/S1973-9087.20.06339-X. Epub 2020 Jul 15. PMID 32667150
- [Background] O'Sullivan O, Barker-Davies RM, Thompson K, Bahadur S, Gough M, Lewis S, Martin M, Segalini A, Wallace G, Phillip R, Cranley M. Rehabilitation post-COVID-19: cross-sectional observations using the Stanford Hall remote assessment tool. BMJ Mil Health. 2023 Jun;169(3):243-248. doi: 10.1136/bmjmilitary-2021-001856. Epub 2021 May 26. PMID 34039689
- [Background] Patel J, Franklin BA, Pujary D, Kaur G, Deodhar A, Kharbanda S, Contractor A. Effects of Supervised Exercise-Based Telerehabilitation on Walk Test Performance and Quality of Life in Patients in India With Chronic Disease: Combatting Covid-19. Int J Telerehabil. 2021 Jun 22;13(1):e6349. doi: 10.5195/ijt.2021.6349. eCollection 2021. PMID 34386155
- [Background] Puterman E, Hives B, Mazara N, Grishin N, Webster J, Hutton S, Koehle MS, Liu Y, Beauchamp MR. COVID-19 Pandemic and Exercise (COPE) trial: a multigroup pragmatic randomised controlled trial examining effects of app-based at-home exercise programs on depressive symptoms. Br J Sports Med. 2022 May;56(10):546-552. doi: 10.1136/bjsports-2021-104379. Epub 2021 Sep 27. PMID 34580067
- [Background] Yang Y, Koenigstorfer J. Determinants of physical activity maintenance during the Covid-19 pandemic: a focus on fitness apps. Transl Behav Med. 2020 Oct 8;10(4):835-842. doi: 10.1093/tbm/ibaa086. PMID 32926160
- [Derived] Salvador-Ruiz AJ, Moral-Munoz JA, Salazar A, Lucena-Anton D, De Sola H, Failde I, Duenas M. Enhancing exercise intervention for patients with post-acute COVID-19 syndrome using mobile health technology: The COVIDReApp randomised controlled trial protocol. Digit Health. 2024 Oct 29;10:20552076241247936. doi: 10.1177/20552076241247936. eCollection 2024 Jan-Dec. PMID 39493634